CLINICAL TRIAL: NCT06672107
Title: Driving Simulator Training to Improve Driving Performance in Veteran Stroke Patients
Brief Title: Driver Training After Stroke
Status: Recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: N5300-R
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: Stroke; Brain injury; Driving; Cognition
MeSH Terms: conditions — Stroke; Brain Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: None Retained — no biospecimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Right hemisphere stroke: Participants with a history of a unilateral stroke affecting the right cerebral hemisphere.
  Interventions: Behavioral: Active Driver Training Intervention; Behavioral: Control Intervention
- Left hemisphere stroke: Participants with a history of a unilateral stroke affecting the left cerebral hemisphere.
  Interventions: Behavioral: Active Driver Training Intervention; Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: Active Driver Training Intervention — simulated driver training focusing on practice of 4 specific driving skills including lane positioning, speed management, collision avoidance, and dashboard attention
  Other Names: Active Training Intervention
Behavioral: Control Intervention — pre-scripted familiarization with driving simulator controls in the absence of any complex driving scenarios, decision making requirements, or feedback pertaining to driving skills

SUMMARY:
One hundred Veteran stroke survivors will participate in both an Active Driver Training intervention and a Control intervention in a fully interactive driving simulator. In addition, all participants will complete pre- and post-intervention driving assessments in the driving simulator to measure driving performance and types of driving errors committed. Half the participants will receive the Active Driver Training first, whereas the other half will receive the Control intervention first. Each Active Driver Training session will provide targeted practice and feedback on each of four unique driving skills including: speed management, collision avoidance, lane positioning, and dashboard attention. The Control intervention will be matched for total time but will only provide extra familiarization with the operation of the driving simulator, with no skill-specific practice. It is predicted that the Active Driver Training Intervention will result in improved driving performance, relative to the Control condition. In addition, after a delay period of at least 6 months, all participants will be re-assessed in the driving simulator and will complete a survey to capture changes in driving status.

DETAILED DESCRIPTION:
In this study, 100 Veteran stroke survivors (half with left hemisphere stroke and half with right hemisphere stroke) will engage in both an Active and a Control simulated driving intervention. The order of interventions (Active first vs. Control first) will be randomly assigned.

Each driving intervention will include weekly training for 3 consecutive weeks, followed by a post-intervention driving assessment. After a 1-week delay, participants will complete the other intervention type (for 3 consecutive weeks) followed by another post-intervention driving assessment. Last, all participants will be re-assessed 6 months later to measure stability of post-intervention driving performance and to complete a questionnaire on current driving status. The driving intervention condition (Active vs. Control) will serve as the main predictor variable in the study.

The Active Driver Training intervention sessions include targeted practice on four critical driving skills, namely, lane positioning, speed management, collision/obstacle avoidance, and dashboard attention. In each driver training session, participants complete all 4 modules sequentially, take a short break, and then repeat the sequence. In other words, participants receive targeted training on each skill six times over the 3-week training period.

In the Control sessions, participants will participate in familiarization drives, for a total duration comparable to the Active Driver Training sessions. The familiarization drive is a pre-programmed feature of the driving simulator that is designed to introduce/familiarize participants with the interactive features of the driving simulator (steering wheel, turn signals, rear-view mirror, etc.) but does not include any complex challenges or situations that require decision-making, and no performance feedback is given.

Simulated driving assessments will be re-administered upon completion of each intervention condition (Active Driver Training vs. Control), and again after a 6-month delay period. The driving assessments involve a challenging drive with multiple speed changes and obstacles and provides an overall score, as well as the number of driving errors committed. Post-intervention Driving Assessment scores will provide an indication of driving improvement due to intervention type, thus serving as the primary outcome variable.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veterans
* History of a unilateral stroke (at least 3 months post-onset)
* Ages 40-80
* pre-morbidly right hand dominant
* prior driving experience/U.S. driver's license

Exclusion Criteria:

* History of other neurologic illness (e.g., TBI, dementia, epilepsy, Parkinson's, etc.)
* History of severe psychiatric illness (e.g., schizophrenia or other psychotic disorders)
* Recent substance abuse/dependence disorder (< 1 year)
* Non-Veteran status

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: U.S. Veteran stroke survivors within the VA Northern California Health Care network
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Driving Score-post Active Training Intervention | 4 weeks
  Numerical score generated from the simulated Driving Assessment that takes place after the Active Driver Training intervention.
Driving Score- post Control Intervention | 4 weeks
  Numerical score generated from the simulated Driving Assessment that takes place after the Control intervention.
6-mo followup Driving Score | 6 months
  Driving Assessment after a 6-mo post-intervention delay

SECONDARY OUTCOMES:
Return to Driving Status-6months | 6 months
  Self reported return to driving status

CONTACTS AND LOCATIONS:
Overall Officials: Krista Schendel Parker, PhD BA, Principal Investigator — VA Northern California Health Care System, Mather, CA
Locations (1):
- VA Northern California Health Care System, Mather, CA, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akinwuntan AE, Wachtel J, Rosen PN. Driving simulation for evaluation and rehabilitation of driving after stroke. J Stroke Cerebrovasc Dis. 2012 Aug;21(6):478-86. doi: 10.1016/j.jstrokecerebrovasdis.2010.12.001. Epub 2011 Jan 14. PMID 21236698
- [Background] Devos H, Akinwuntan AE, Nieuwboer A, Truijen S, Tant M, De Weerdt W. Screening for fitness to drive after stroke: a systematic review and meta-analysis. Neurology. 2011 Feb 22;76(8):747-56. doi: 10.1212/WNL.0b013e31820d6300. PMID 21339502
- [Background] Akinwuntan AE, Devos H, Verheyden G, Baten G, Kiekens C, Feys H, De Weerdt W. Retraining moderately impaired stroke survivors in driving-related visual attention skills. Top Stroke Rehabil. 2010 Sep-Oct;17(5):328-36. doi: 10.1310/tsr1705-328. PMID 21131257
- [Background] Perrier MJ, Korner-Bitensky N, Petzold A, Mayo N. The risk of motor vehicle crashes and traffic citations post stroke: a structured review. Top Stroke Rehabil. 2010 May-Jun;17(3):191-6. doi: 10.1310/tsr1703-191. PMID 20797963